CLINICAL TRIAL: NCT00120796
Title: Lamivudine and Therapeutic Vaccine Evaluation in Senegalese Patients With Chronic Hepatitis B Infection
Brief Title: Lamivudine and Therapeutic Vaccine Evaluation in Senegalese Patients With Chronic Hepatitis B Infection (ANRS 12100 HEPADAK-2)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: poor patient recrutment
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Director, ANRS
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 12100 HEPADAK-2
Record Dates: First submitted 2005-07-12; First posted 2005-07-19 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2008-03

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Hepatitis B Vaccines; Lamivudine
MeSH Terms: conditions — Hepatitis B | interventions — Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Lamivudine alone
  Interventions: Drug: Lamivudine
- 2 (Experimental): Lamivudine + Vaccine
  Interventions: Drug: Lamivudine; Biological: Recombinant hepatitis B surface antigen

INTERVENTIONS:
Drug: Lamivudine
Biological: Recombinant hepatitis B surface antigen
  Arms: 2

SUMMARY:
Chronic hepatitis B infection is a major public health issue in Senegal. The study will compare the efficacy of the treatment strategy combining Lamivudine and therapeutic vaccine (12 intra-muscular injections over a 6-month period) to a treatment with Lamivudine alone on the control of viral replication in patients with a replicative hepatitis B virus (HBV) infection and an increase in hepatic enzymes.

DETAILED DESCRIPTION:
Hepatitis B infection with a prevalence higher than 15% of positive Ag HBs subjects is a major public health issue in Senegal. A program of treatment of patients presenting with hepatic disease is currently ongoing through a network of specialists in GI tract and liver diseases. Hepatitis B is a real threat in the Senegalese population as showed in a pilot study (HEPADAK I) performed at the Dakar Hospital Principal (DHP) in Dakar among 100 blood donors and 50 patients with liver disease. This study allowed us to better characterize the strains at the molecular level. The aim of the project is to assess a pragmatic treatment strategy which can be applied to Senegal or other developing countries for patients requiring treatment. A recent Japanese study performed in Ag HBe positive patients reported the interest of the combination of Lamivudine (LAM) and a therapeutic vaccine with the negativation of viral load in 100% of patients after one year of treatment. It is important to show that such a treatment with 12 intra-muscular injections of the vaccine over a 6-month period is feasible in Africa and to assess the results of such a treatment in the Senegalese population, which is mainly AgHBe negative.

The study HEPADAK 2 is a randomized open label study which will compare the efficacy of the treatment strategy combining Lamivudine and therapeutic vaccine (12 intra-muscular injections of Engerix B over a 6-month period) to a treatment with Lamivudine alone on the control of viral replication in patients with a replicative HBV infection and an increase in transaminases.

Eligible patients have to be HIV, HDV and HCV negative and will have to i) give their written informed consent; ii) have a B hepatitis grade over or equal to F2 with the Metavir score, DNA HBV greater than 105 copies/mL (or 104 copies/mL if Ag Hbe -) , ALAT greater than 1.3 times the upper limit of the normal; iii) accept to have a liver biopsy and to be followed for this protocol at the DHP. After a 3-month treatment with Lamivudine, patients whose viral load is negative or at least decreased by 4 Log will be randomized to the same treatment for a further 9-month period or to the same treatment combined with 12 injections of vaccine over 6 months. The main endpoints are undetectability of HBV DNA blood level 12 months after treatment initiation and 6 months after the end of the treatment. Secondary endpoints will be HBV DNA blood levels at 3, 6, 9 and 12 months after the end of the treatment, transaminases blood level, Lamivudine treatment compliance, the feasibility of the vaccine injections schedule, safety, AgHBe seroconversion (in positive patients) and negativation of AgHBs. Two hundred ten patients have to be included (70 in the Lamivudine group, and 140 in the Lamivudine + vaccine group) in order to show a difference of at least 20% in the percentage of patients with an undetectable viral load at 12 months (70% expected under Lamivudine monotherapy), with a power of 90%, an alpha risk equal to 5% and a bilateral test. Patients with a virological failure will be maintained or retreated with Lamivudine. For the patients with an YMDD mutation, a treatment with Adefovir Dipivoxil will be possible. Patients' inclusion is planned to start in January 2005 and end after 12 or 18 months. Patients will be treated during one year and followed one year without treatment in the study protocol, and then will be managed if necessary

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Liver biopsy acceptation
* B hepatitis grade over or equal to F2 Metavir score
* DNA HBV greater than 100000 copies/mL (or 10000 copies/mL if Ag Hbe negative)
* ALAT greater than 1.3 times the upper normal limit

Exclusion Criteria:

* HCV, HDV and HIV positive
* Pregnancy
* Decompensated liver cirrhosis
* Pretreated patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
undetectability of HBV DNA blood level | 12 months after treatment initiation (6 months after the end of the treatment)

SECONDARY OUTCOMES:
HBV DNA blood levels | 3, 6, 9 and 12 months after the end of the treatment
Transaminases blood level | 12 months
Lamivudine treatment compliance | 12 months
Feasibility of the vaccine injections schedule | 6 months
Safety | 12 months
AgHBe seroconversion (in positive patients) | 12 months
AgHBs negativation | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Papa Saliou Mbaye, Principal Investigator — Hopital Principal de Dakar Senegal; Muriel Vray, Study Chair — Institut Pasteur, Paris France
Locations (1):
- Hopital Principal, Dakar, Senegal